CLINICAL TRIAL: NCT06351995
Title: Neostigmine and Glycopyrrolate by Iontophoresis to Induce Bowel Evacuation
Brief Title: Neostigmine and Glycopyrrolate by Iontophoresis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chris Cardozo, Principal Investigator, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOR-19-22
Record Dates: First submitted 2024-03-21; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Constipation; Fecal Incontinence; Neurogenic Bowel
Keywords: Neostigmine; Glycopyrrolate; Transdermal; Intravenous; Pharmacokinetic; Constipation; Bowel Control; Mass Spectroscopy; Stool Incontinence
MeSH Terms: conditions — Spinal Cord Injuries; Constipation; Fecal Incontinence; Neurogenic Bowel; Encopresis | interventions — Glycopyrrolate; Iontophoresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Primary (Experimental): Subjects will receive medication administration intravenously, then through a wired ION system of NEO + GEO.
  Interventions: Drug: Combination of Neostigmine and Glycopyrrolate; Device: I-Box by Dynatronics

INTERVENTIONS:
Drug: Combination of Neostigmine and Glycopyrrolate — Intravenous or transdermal
Device: I-Box by Dynatronics — Electric field conducting drugs through the skin without compromising its integrity
  Other Names: Iontophoresis

SUMMARY:
To determine a lower effective dose of neostigmine to induce bowel evacuation by transcutaneous administration by iontophoresis.

DETAILED DESCRIPTION:
Subjects will progress to receive the standard dose previously reported and employed for these agents [NEO (0.07 mg/kg) + GLY (0.014 mg/kg)] by transdermal administration by use of a wired ION system. NEO and GLY can be delivered into the systemic circulation by transcutaneous route by ION to induce a safe and predictable bowel evacuation in persons with SCI. If digital rectal stimulation was utilized in the screening session, this method will be utilized for the remaining sessions as needed at the discretion of the primary investigator. In the anesthesiology literature, a ratio of NEO to GLY of about 5 to 1 has been employed in clinical situations. Participants will be requested not to have bowel care for at least 1 day prior to the study. The subject will assume normal bowel evacuation position until a bowel movement occurs. Privacy draping and privacy will be provided at the time of bowel evacuation. The subjects will be monitored for 120 minutes. A minimum of two research personnel will be present during the study visit to record all of data and perform the tasks required.

From recent work, it is extrapolated that 85 to 90% of participants will have a bowel evacuation to transdermal administration of NEO by ION. The pharmacokinetics of only those who have a bowel evacuation to NEO will be used in the calculation to determine the peak plasma concentration (PPC) and area under the curve (AUC) of NEO and GLY. The PPC and AUC for the non-responders to NEO will be analyzed separately; it is speculated that the PPC of NEO for the non-responders will be blunted-that is, at least below the mean value of the PPC for NEO administration.

The absorption of study agents is, to a certain extent, subject-specific because of differential absorption through the skin. As such, each participant is expected to display differing responses: shorter or longer times to bowel evacuation (or the absence of bowel evacuation), as well as the absence or presence of cholinergic (increased bowel activity, bradycardia, bronchoconstriction) or anti-cholinergic activity, as previously described in the text above. The pharmacokinetic data will, to a large extent, reflect this variability in transdermal drug absorption. The data collected will include the presence or absence of bowel evacuation, time to bowel evacuation, consistency (Bristol stool scale), and quantity (by weight). The presence/number of cholinergic and anti-cholinergic side-effects on a standardized point scale will be determined, as well as their severity (e.g., mild, moderate, or severe). Heart rate, blood pressure, oxygen saturation, and pulmonary mechanics (airway patency by impulse oscillation system) will be recorded at baseline and sequentially at intervals the initiation of ION (at 5, 10, 15, 20, 30, 45, 60, 90, and 120 minutes).

To quantitate the amount of these agents absorbed into the systemic circulation, pharmacokinetic studies will be performed for 2 hours after the start of transdermal drug delivery. Venous blood (2 ml) will be collected into an EDTA tube for both agents at the following time points: baseline (time zero), 5, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, 360, and 480 minutes. Upon drawing, the blood will be placed in an ice bath and spun using a centrifuge within 5 minutes of collection. Upon completion of 5 minutes of centrifugation, the plasma will be aliquoted into two separate vials, with equal volumes and labeled with date and time of draw, study information, NEO or GLY testing destination, and the subject's unique identifier. The transfer vials will be inserted into dry ice for at least 10 minutes, after which they will be placed into the -80 degrees Celsius freezer. Plasma levels of NEO and of GLY will be batched and measured at a later date. A file designating the tubes with random numbers associated with the draw times will be created for each subject to conceal the sequence of draw and to attempt the removal of possible bias during the measurement and recording of the concentrations of NEO and GLY. NEO and GLY will be measured by mass spectroscopy.

To determine the reproducibility of the transdermal absorption of NEO and GLY, as well as the potential side-effects, subjects will again receive NEO (0.07 mg/kg) + GLY (0.014 mg/kg) by transdermal administration by use of a wired ION system. Additionally, digital rectal stimulation will be utilized as needed at the discretion of the primary investigator. Pharmacokinetic data and all other measurements and questionnaires that were previously obtained will be acquired once again and compared to Trial 1.

The investigators will have obtained pharmacokinetic data on each participant from Study 1. From the data acquired, the peak plasma concentration (PPC) and the area under the curve (AUC) for NEO will be calculated. The hypothesis is that the PPC for NEO will correlate more closely with bowel evacuation than its AUC, and the AUC for GLY will correlate more closely with anti-cholinergic symptoms than its PPC, but this prediction is just speculation prior to obtaining and analyzing the data. If the plasma concentration of each NEO and GLY are solely responsible for determining biological effects (e.g., cholinergic and anti-cholinergic), then the investigators would predict that there will be a direct and strong correlation of drug levels with those endpoints. However, if the biological effects are primary determined by end-organ responsiveness, then the correlation between drug concentration and observed endpoints will be tenuous, at best. If both plasma concentration and end-organ responsiveness play a role in bowel evacuation and cholinergic side-effect, then an effect of plasma concentrations will still be evident, but not as strong.

Determination of a Lower Effective Dose of NEO to Induce Bowel Evacuation Because 85-90% of participants are anticipated to have a bowel evacuation from NEO administration at the dose previously employed (standard dose: NEO 0.07 mg/kg), the dose administered is most probably well above the lowest effective dose to achieve the biological desired effect ("ceiling effect"). If the lowest effective dose can be determined, side-effects from NEO administration will be reduced. As such, to identify the upper limit of the lowest effective dose, the dose of NEO will be titrated down until the effect on the primary end organ is lost-that is, until bowel evacuation no longer occurs after drug administration in at least 50% of the participants. Thus, to determine if a lower dose of NEO will still result in bowel evacuation, participants will have the dose of NEO reduced by 25% (with the dose of GLY also reduced by 25%). The total volume of the drugs applied to the patch will be kept constant. In these dose reduction experiments, pharmacokinetic data (e.g., AUC and PPC) will be obtained on each participant for each reduction in dose of NEO. All other measurements and questionnaires that were obtained in Study 1 will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 18 to 89;
* Chronic SCI (>1 year post injury);
* You have documented constipation/difficulty with bowel evacuation and/or experience pain, straining, or fecal incontinence.

Exclusion Criteria:

* Previous adverse reaction or hypersensitivity to electrical stimulation;
* Known sensitivity (prior reaction or allergy) to neostigmine or glycopyrrolate
* History of mechanical obstruction (physical blockage) of the GI or urinary tract (e.g., due to scar tissues forming after surgery, gallstones);
* Myocardial infarction (heart attack) within 6 months of trial;
* Malignant and/or uncontrollable hypertension (high blood pressure), defined as a blood pressure reading of 160/100 mmHg or higher with or without taking 3 or more different classes of anti-hypertensive medications (drugs used to treat high blood pressure);
* Organ damage (heart & kidney) and/or transient ischemic attack/cerebrovascular accident (TIA-CVA, or stroke) as a result of hypertension;
* Known past history of coronary artery disease or bradyarrhythmia (slow heart rate);
* Symptomatic orthostatic hypotension (low blood pressure with possible dizziness/fainting);
* Deep brain stimulation;
* Pregnancy (women who are sexually active and of childbearing potential must utilize a method of contraception and agree to maintain a contraceptive method until completion of the study);
* Lactating, nursing females;
* Inability to provide informed consent determined by Montreal Cognitive Assessment Test (MoCA) score of 20 or less. This test is used to detect mild cognitive impairment;
* History of ingrown hair folliculitis (inflammation of hair follicles)
* Concurrent illness (with or without fever), such as lower respiratory illnesses, increased mucous/secretin production, congestive heart failure (CHF), or pneumonia;
* Currently taking the following medications: Bethanechol, Chloroquine, Colistin, Penicillamine, Lithium, Methylcellulose, Trimeprazine, Verapamil, Phenothiazines, Sparfloxacin, Amitriptyline, Doxepin, Imipramine, Potassium chloride, Saquinavir, Dronedarone, Cisapride, Bepridil, Terfenadine, Amiodarone, Ziprasidone, or any medication(s) that could result in adverse reactions with neostigmine and/or glycopyrrolate, as determined by a study physician;
* Currently taking cholinesterase inhibitors, such as those for Parkinson's Disease (PD) or dementia (rivastigmine, donepezil etc.), or medication with anticholinergic activity, such as anti-depressants;
* Myasthenia gravis;
* EKG abnormalities such as bradycardia, prolonged QTc interval, axis shift, bundle branch block, Wolff-Parkinson-White Syndrome (WPW syndrome), 2nd and 3rd degree heart blocks etc. (determined at screening 12-lead EKG);
* Chronic gastrointestinal (GI) disease such as inflammatory bowel disease (IBD), irritable bowel syndrome with constipation (IBS-C), or other causes of difficulty with stool evacuation such as hypothyroidism (underactive thyroid);
* Fever (as an isolated symptom without "illness"), or who may be exposed to high environmental temperatures
* Concurrent participation in a research study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of bowel evacuation | Up to 2 hours post Neostigmine and Glycopyrrolate administration
  Presence or absence of bowel evacuation post Neostigmine and Glycopyrrolate administration
Time to bowel evacuation | Up to 2 hours post Neostigmine and Glycopyrrolate administration
  Time to bowel evacuation post Neostigmine and Glycopyrrolate administration
Stool Consistency | Up to 2 hours post Neostigmine and Glycopyrrolate administration
  Stool Consistency (Bristol stool scale) post bowel evacuation
Stool Quantity | Up to 2 hours post Neostigmine and Glycopyrrolate administration
  Stool quantity (by weight) post bowel evacuation

SECONDARY OUTCOMES:
Presence or absence of headache, dry mouth, muscle twitching and abdominal cramps. | Up to 2 hours post Neostigmine and Glycopyrrolate administration
  The presence/number of cholinergic and anti-cholinergic side-effects on a standardized point scale will be determined, as well as their severity (e.g., mild, moderate, or severe).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Cardozo, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No